CLINICAL TRIAL: NCT01649934
Title: The Use of Implementation Intentions to Increase the Appointment Attendance of Operation Enduring Freedom/Operation Iraqi Freedom (OEF/OIF) Veterans
Brief Title: The Use of Implementation Intentions to Increase the Appointment Attendance of OEF/OIF Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 01634
Record Dates: First submitted 2012-07-22; First posted 2012-07-25 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Brain Injuries
Keywords: Appointments and Schedules
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Scheduling as Usual (No Intervention): Participants will be subject to the current appointment scheduling procedures.
- Contact Clinic (Experimental): This group will be required to contact the clinic themselves to make appointments.
  Interventions: Behavioral: Contact Clinic
- Implementation Intentions (Experimental): This group will create Implementation Intentions to contact the clinic to make their appointments and to attend those appointments.
  Interventions: Behavioral: Implementation Intention

INTERVENTIONS:
Behavioral: Implementation Intention — Implementation Intentions are a series of what/when/where statements that a participant will make to create automatic cues to complete a behaviorally advantageous action.
  Arms: Implementation Intentions
Behavioral: Contact Clinic — Participants will be asked to sign a form indicating their need to contact the recommended clinics to make their appointments.
  Arms: Contact Clinic

SUMMARY:
The purpose of the current pilot study will be to utilize implementation intentions to increase patient compliance with appointment attendance. Participants in the current study will be individuals referred for evaluation of their treatment needs. Experimental groups will create a simple induction consisting of "what/when/where" statements (implementation intentions) with the intention of increasing their rate of calling to schedule and subsequently attend appointments associated with their care. It is anticipated that participants who take an active role in their plan and utilize the implementation intention procedures will be more likely to make and attend the appointments suggested by their treating clinician. This pilot project will provide valuable initial data as to the potential effectiveness of a simple, cost-effective means of increasing appointment attendance. If successful, it could lead to cost savings and a decrease in the appointment wait time for people by increasing the utilization of available appointments.

DETAILED DESCRIPTION:
The purpose of the current pilot study will be to utilize implementation intentions to increase patient compliance with appointment attendance. It is anticipated that participants who take an active role in their plan and utilize the implementation intention procedures will be more likely to make and attend the appointments suggested by their treating clinician. Sixty participants will be recruited to participate in the research project. Participants in the current study will be individuals referred for a secondary Traumatic Brain Injury (TBI) screen. This appointment serves to develop the plan of care that will be used for determination of the treatments that would be beneficial to the Veteran and as such the appointments necessary for further assessment or treatment in affiliated clinics (i.e. mental health, physical therapy, neuropsychology). Twenty participants will serve as controls who will receive treatment planning as usual. Twenty participants will receive treatment as usual but will be asked to contact the clinics directly to make their appointments. Twenty participants will be provided with a simple implementation intention induction. The simple induction will consist of the creation of "what/when/where" statements surrounding their intention to call to schedule and to attend medical appointments associated with their care. Research staff will then monitor the participants' appointment schedule daily to determine if they made the appropriate appointments and subsequently attended those appointments. Primary data for the examination will be these yes/no data points as to whether the participant successfully adhered to their initial intention to schedule the prescribed appointments. Additionally, for those who schedule the prescribed appointments, the latency in days from the time they indicated they intended to make their appointments will serve as a measure of their compliance. Across all groups, attendance at those appointments will be recorded to determine if the procedures lead to an increase in their attendance at their appointments compared to the treatment as usual group. This pilot project will provide valuable initial data as to the potential effectiveness of a simple, cost-effective means of increasing appointment attendance. If successful, it could lead to cost savings to the VA system and a decrease in the appointment wait time for Veterans by increasing the utilization of available appointments.

ELIGIBILITY:
Inclusion Criteria:

* Completed appointment for secondary TBI screen
* English speaker

Exclusion Criteria:

* Neurological injury leading to dementia
* In ability to consent owing to cognitive barriers
* Non-English speaker
* Unable to schedule appointments the next working day after their secondary screen

Ages: 22 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2013-06; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Attendance at Scheduled Appointments | Over a 60 Day Period
  The attendance of the participants at their scheduled appointments will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph F Kulas, Ph.D., Principal Investigator — VA Connecticut Healthcare System
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sheeran P, Orbell S. Using implementation intentions to increase attendance for cervical cancer screening. Health Psychol. 2000 May;19(3):283-9. doi: 10.1037//0278-6133.19.3.283. PMID 10868773
- [Background] Collins J, Santamaria N, Clayton L. Why outpatients fail to attend their scheduled appointments: a prospective comparison of differences between attenders and non-attenders. Aust Health Rev. 2003;26(1):52-63. doi: 10.1071/ah030052. PMID 15485374
- [Background] Thornton R, Ballard K. Why military personnel fail to keep medical appointments. J R Army Med Corps. 2008 Mar;154(1):26-30. doi: 10.1136/jramc-154-01-08. PMID 19090383
- [Background] Stiggelbout AM, Van der Weijden T, De Wit MP, Frosch D, Legare F, Montori VM, Trevena L, Elwyn G. Shared decision making: really putting patients at the centre of healthcare. BMJ. 2012 Jan 27;344:e256. doi: 10.1136/bmj.e256. PMID 22286508
- [Background] Guy R, Hocking J, Wand H, Stott S, Ali H, Kaldor J. How effective are short message service reminders at increasing clinic attendance? A meta-analysis and systematic review. Health Serv Res. 2012 Apr;47(2):614-32. doi: 10.1111/j.1475-6773.2011.01342.x. Epub 2011 Nov 8. PMID 22091980
- [Background] O'Carroll R, Dennis M, Johnston M, Sudlow C. Improving adherence to medication in stroke survivors (IAMSS): a randomised controlled trial: study protocol. BMC Neurol. 2010 Feb 24;10:15. doi: 10.1186/1471-2377-10-15. PMID 20181255
- [Background] Sheeran P, Aubrey R, Kellett S. Increasing attendance for psychotherapy: implementation intentions and the self-regulation of attendance-related negative affect. J Consult Clin Psychol. 2007 Dec;75(6):853-63. doi: 10.1037/0022-006X.75.6.853. PMID 18085903
- [Background] Brown I, Sheeran P, Reuber M. Enhancing antiepileptic drug adherence: a randomized controlled trial. Epilepsy Behav. 2009 Dec;16(4):634-9. doi: 10.1016/j.yebeh.2009.09.014. Epub 2009 Oct 27. PMID 19864187
- [Background] Milkman KL, Beshears J, Choi JJ, Laibson D, Madrian BC. Using implementation intentions prompts to enhance influenza vaccination rates. Proc Natl Acad Sci U S A. 2011 Jun 28;108(26):10415-20. doi: 10.1073/pnas.1103170108. Epub 2011 Jun 13. PMID 21670283